CLINICAL TRIAL: NCT03596814
Title: Retrospective and Descriptive Analysis of the Regimens of Treatment With FVIII, FIX and By-passing Agents for Hemophiliacs A or B With or Without Inhibitors, From the Existing Registry BERHLINGO, Before and After the Launch of New Entended Half-life Clotting Factors in Seven Haemophilia Treatment Centers in France
Brief Title: MOTHIF II : THERAPEUTIC MANAGEMENT AND USE OF CLOTTING FACTORS IN HEMOPHILIA A & B IN FRANCE II
Acronym: MOTHIF II
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0288
Record Dates: First submitted 2018-03-22; First posted 2018-07-24 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia
Keywords: Hemophilia A; Hemophilia B; Research database; Clotting Factors; Regimen of Treatment; Impact Budget Analysis
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Interventional study — Retrospective data

SUMMARY:
MOTHIF II is a non-interventional, multicenter, retrospective, observational data collection in seven French Haemophilia Treatment Centers of the BERHLINGO network. In the context of the arrival of new extended half-life products, the MOTHIF II study aims to describe the changes in therapeutic management of patients with hemophilia A & B, following the provision of FVIII and FIX extended half-life factors in France; it will also permit to carry out a budget impact analysis to quantify the economic significance of this new era.

DETAILED DESCRIPTION:
Treatment regimens for haemophiliacs patients treated with clotting factors will be analysed globally for the patients of the two periods, by subgroup:

* type of hemophilia: A or B
* severity: severe, moderate, mild
* history of inhibitors

and then for each subgroup:

* by regimen: 1) Prophylaxis 2) On demand 3) ITI
* by type of clotting factors: FVIII or FIX or by-passing agents, plasma-derived or recombinant, standard or extended half-life clotting factors, INN

Will also be included in the analyse:

* demographic data: age (years)
* clinical data: weight (kgs) if available
* treatment data: regimen, consumptions (number of UI of clotting factors consumed on the period) and costs of clotting factors (€).

ELIGIBILITY:
Inclusion Criteria:

* All patients hemophiliac A or B, with or without inhibitors, included in the Nhemo (7 centres) and the Behrlingo database, treated with factor 8 or factor 9 products or by-passing agents
* All Hemophilia A or B patients of any severity without inhibitors, included in the NHEMO database and the BEHRLINGO database, without any treatment by clotting factors
* All Hemophilia A or B patients having given consent to be included in the study (2 times 12 months), during their usual follow-up (consultation…). For the other patients, a derogation from the obligation to inform the patients will be made to the CNIL.

Exclusion Criteria:

* patients under guardianship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Estimation of the population of the study: 2 000 patients will be enrolled by seven centers in France (treated or not).
  Settings : 7 Hemophilia Traitement Center of Western France : Angers, Brest, Caen, Le Mans, Nantes, Rennes and Tours
Sampling Method: Non-Probability Sample
Enrollment: 2072 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
A comparison of the consumptions of CF before and after the laucnh of EHL CF is an assessment of the the impact of EHL CF on the treatment of haemophiliacs patients | 24 months (1st July 2015- 30th June 2016 & 1st July 2017-30th June 2018 (before and after the launch of extended half-life CF in France))
  Deletion of the measure of % of switch

CONTACTS AND LOCATIONS:
Overall Officials: Marc TROSSAERT, Dr, Principal Investigator — Nantes University Hospital
Locations (7):
- France (7):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Caen university Hospital, Caen
  - Le Mans University Hospital, Le Mans
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours